CLINICAL TRIAL: NCT03593850
Title: Music for the Management of Pain in Primary Dysmenorrhea in Students of the School of Medicine and Health Sciences From the Universidad Del Rosario
Brief Title: Music for Pain in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Rosario (Other)
Responsible Party: Principal Investigator, Juan S. Martin-Saavedra, Research Assistant, Universidad del Rosario
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEI856
Record Dates: First submitted 2018-06-04; First posted 2018-07-20 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Pain, Menstrual; Primary Dysmenorrhea
Keywords: Pain management; Pain; Primary dysmenorrhea; Music; Music Therapy
MeSH Terms: conditions — Dysmenorrhea; Agnosia; Pain | interventions — SIR1 protein, S cerevisiae

STUDY DESIGN:
Intervention Model Description: Single blinded, two parallel group, randomized clinical trial. The experimental group received listen to a son composed exclusively for this trial while control group rested for the same amount of time in silence.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Computer block randomization was used to generate allocation sequence of codes. Allocation was done on the same day of the intervention, patients were given opaque envelope according to the randomization codes. The envelop contained instructions to access the allocated intervention. After baseline data collection patients entered the intervention room and opened the envelop inside while investigator waited outside. Both patients had headphones on and used the same device to access the intervention assuring blinding of the investigator. After the intervention ended, patient closed the intervention file and account to the intervention. All patients were instructed to nor reveal or comment anything about the intervention at any time after the intervention was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music group (Experimental): Patients in this arm listened through headphones to a song of 29 minutes and 32 seconds duration. The song was composed entirely by investigator Juan Martin-Saavedra and registered to copyright and authorship regulatory entities from Colombia under the name "Occasio adolore" (Musical piece No. 5-559-355 and Phonogram No. 12-105-295 of Colombia's Copyright authorship agency). Patients were instructed to avoid using cellphones or other activities during the time of the intervention. Patients receive the intervention in the same room as the Silence group, but for the intervention they were always alone. The room was located in a low transit place with low ambient noise.
  Interventions: Behavioral: Music group
- Silence group (Active Comparator): Patients on the silence group listened to a 29 minute and 32 second audio file that produced no sounds with headphones on. Patients were instructed to avoid using cellphones or other activities during the time of the intervention. Patients receive the intervention in the same room as the Music group, but for the intervention they were always alone. The room was located in a low transit place with low ambient noise.
  Interventions: Behavioral: Silence Group

INTERVENTIONS:
Behavioral: Music group — The song was composed on a C major scale and a 60 bpm tempo. The song was composed with high consonance using simple melodic progressions on the C major scale, and using natural positions for chords. No percussion or lyrics were used for the song, and the following instruments were used in the composition: electric guitar and keyboards, violin (digital), cello (digital), clarinet (digital), synthesizers (digital), and fretless bass (digital).
  Other Names: Occasio adolore
  Arms: Music group
Behavioral: Silence Group — Audio file that contained no sounds.
  Other Names: Silence
  Arms: Silence group

SUMMARY:
Primary dysmenorrhea is defined as lower abdominal pain that occurs during menses and is not secondary to any type of pelvic disease. It is considered the most common condition in reproductive age women. First line of treatment are non-steroidal anti-inflammatory drugs (NSAIDS), or oral contraceptives (OCC). This two forms of treatment have not demonstrated 100% efficacy, and adverse events and contraindications for both exist. Moreover, studies have demonstrated that an important women do not use, or don't like to use, pharmacological treatment. Music have demonstrated analgesic effects in different clinical contexts, and has emerged as an important form of complementary therapy in the management of pain. To the researcher's knowledge, no studies have been conducted to evaluate music's effectiveness in pain secondary to primary dysmenorrhea.

The following is the protocol for a randomized, single blinded, clinical trial, where an experimental group listened to a 30 minute song, and was compared to a control group that rest in silence for the same time and conditions. It was expected that music will produce a larger, and significant, effect on pain reduction when compared to the control silence group according to pain measured through a 10 cm Visual Analogue Scale (VAS) in young women from the School of Medicine and Health Sciences at the Universidad del Rosario, Bogota DC, Colombia. Additionally, the investigators wanted to evaluate the clinical effect of music and analgesic requirements, anxiety and vital signs were also measured.

DETAILED DESCRIPTION:
Primary Dysmenorrhea (PD) is defined as pain in the lower abdomen, that occurs always during menses, in the absence of pelvic pathology, and lasts about 24-72 hours. It initiates during the first 24 months after menarche. Other symptoms like, emotional lability, anxiety, nausea, headache, and others may accompany the pain. It is considered the most common condition of reproductive age women, and is considered one of the most important causes for school or work absence in this population.

Music has been proposed as a complementary therapy for the management of pain, and a large body of clinical evidence supports its use on clinical context. Additionally, functional imaging research has found that music activates areas related to pain modulation and perception like the periaqueductal gray matter. Moreover music seems to modify brain activity during pain perception. Music has been shown to be effective in relieving pain secondary to surgery, in cancer related pain, and other types of pain, but it has not been studied for primary dysmenorrhea.

This randomized clinical trial was designed with the following objectives

General Objective: To evaluate the efficacy of music listening, compared to a control group that rested in silence, in the painful experience secondary to primary dysmenorrhea in women of 18 years or older from the School of Medicine and Health Sciences at the Universidad del Rosario, Bogotá DC., Colombia.

Specific Objectives:

1. Description of demographic data, clinical, gynecological, and obstetric background from the study population.
2. Description of pain management, secondary to PD, used by the study population.
3. Evaluate the usual pain secondary to PD, as reported by the study participants through a Visual Analogue Scale (VAS)
4. To explore if the acute perception of pain secondary to PD, as reported by participants using a VAS, before the intervention, is different between the study groups.
5. To evaluate if the acute perception of pain secondary to PD, as reported by participants using a VAS, after the intervention, differs between those that listened to music and those that rested in silence.
6. To explore if a difference in the reduction of pain, as reported by participants using a VAS, from the moment before to the moment after the intervention exists between those in the music group compared to those in the silence group.
7. To evaluate if the acute perception of pain secondary to PD, as reported by participants using a VAS, 3-6 hours after the intervention, differs between those that listened to music and those that rested in silence.
8. To evaluate if the anxiety secondary to PD, as reported by participants using a validated Spanish short version of the Zung scale, differs between groups, before and after the intervention.
9. To evaluate if a difference in the reported requirements of analgesic drugs is different between the study groups after and 3-6 hours after the intervention.
10. To evaluate if a difference in heart rate, systolic and diastolic blood pressure is identified between groups, using a previously calibrated digital sphyngmomanometer.

The investigators hypothesized that listening to an instrumental song, unknown to the patient, will have a significant effect on pain relief. Additionally, investigators hypothesized that music listening will have a clinical effect big enough to also impact analgesic requirements and anxiety scores .

Primary endpoint was pain reduction from the moment before to after the intervention. Pain reduction is the better way to evaluate analgesia efficacy and was the proper approach for these protocol's main objective, which was efficacy of music on pain relief secondary to primary dysmenorrhea.

For achieving these aims and answering research questions, a randomized clinical trial was designed. As patients can't be blinded from listening or not to music, a single blinded approach was decided. Furthermore, methodology for recruitment was designed to blind patients from allocation until the day of the intervention and a speech was used to avoid patients to identify the primary endpoint. Additionally, patients were explained that two interventions were used, but it was not specified that silence group was the control group, to assure proper blinding and avoid further bias of results. Silence was decided as a control intervention as comparison with drug placebo may not be adequate due to differences in the types of intervention.

To isolate the music effects the investigators decided on using a completely new and unknown song. The song was planned and composed exclusively for the research, so all patients allocated to the music group listened to the exact same musical piece.

ELIGIBILITY:
Inclusion Criteria:

* Legal and cognitive capacity for informed consent.
* Suffering from primary dysmenorrhea (low abdominal pain associated to menses).
* Being able to understand and use the measuring tools and questionnaires.

Exclusion Criteria:

* Previous diagnosis of pelvic pathology.
* Diagnosis of hearing impairment.
* Diagnosis of neurologic or endocrinological disease.
* Psychiatric condition diagnosed.
* Known or reported previous substance abuse.
* Current use of psychiatric drugs.
* Cancer diagnosis
* Diagnosed diabetes mellitus or heart disease.
* Previous advance musical training (defined as any form of music training in addition to that received during normal school classes).
* Irregular menstrual cycles.
* Previous pregnancy.
* Current use or use of any hormonal contraceptive therapy in the last 2 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 649 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan S Martin-Saavedra, MD, Principal Investigator — Universidad del Rosario; Angela M Ruiz-Sternberg, MD, MSc, Study Director — Universidad del Rosario
Locations (1):
- Escuela de Medicina y Ciencias de la Salud- Universidad del Rosario, Bogotá, Capital District, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Results fromt the research will be made available as supplemental data or digital content published with the final manuscript. Additional information like the study protocol, statistic analysis plan performed, and copy of the informed consent will be available by request to the email: juans.martin@urosario.edu.co
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Complete database will be made available with publication of the manuscript. Other information will be accessible by request to the email: juans.martin@urosario.edu.co
Access Criteria: Complete database results will be available as digital content with the final manuscript. Additional data will be given by request by email and requester will require to send a letter with signature stating the reason for requesting additional information.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited and between September 2017 to April 2018 from the School of Medicine and Health Sciences, and the School of Mathematics and Natural Sciences from Universidad del Rosario. Assessment, data collection, and intervention occurred within the facilities of the School of Medicine and Health Sciences from Universidad del Rosario, Bogota D.C., Colombia.
Pre-assignment Details: A total of 597 participants were excluded: 470 did not met inclusion criteria, 98 declined to participate, and 29 signed consent but never came for randomization and the intervention.
Period: Primary Endpoint
Arm/Group | Music Group | Silence Group
Started | 29 | 23
Received Allocated Intervention and Completed Post-intervention Outcomes (Primary Endpoint) | 29 | 23 (1 patient took analgesics and did not disclose it prior to completing the allocated intervention)
Completed | 29 (Included in primary endpoint analysis) | 22 (Included in primary endpoint analysis (Intention to treat))
Not Completed | 0 | 1
Period: 3-6 Hours Post Intervention Outcomes
Arm/Group | Music Group | Silence Group
Started | 29 | 22
Completed (Completed and returned 3-6 hours post-intervention outcome questionnaires) | 27 | 19
Not Completed | 2 | 3
Not completed — Did not returned or filled wrongly the outcome questionnaire | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Music Group | Silence Group | Total
Number analyzed (Participants) | 29 | 23 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.1 (2.27) | 19.57 (1.31) | 19.87 (1.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 23 | 52
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Colombia | 29 | 23 | 52
University program [Count of Participants; unit: Participants]
  Medicine | 6 | 10 | 16
  Phonoaudiology | 5 | 7 | 12
  Physiotherapy | 8 | 4 | 12
  Psychology | 5 | 2 | 7
  Other (Epidemiology, Gynecology, Biology) | 5 | 0 | 5
Academic semester [Count of Participants; unit: Participants]
  First to Fifth | 21 | 15 | 36
  Sixth to Tenth | 8 | 8 | 16
Presence of comorbidities [Count of Participants; unit: Participants]
  Yes | 4 | 3 | 7
  No | 25 | 20 | 45
History of surgeries in their lifetime [Count of Participants; unit: Participants]
  Yes | 9 | 6 | 15
  No | 20 | 17 | 37
Age at menarche [Mean (Standard Deviation); unit: years] | 12.14 (1.51) | 12.17 (1.11) | 12.15 (1.33)
Intermenstrual time [Mean (Standard Deviation); unit: days] | 29.07 (2.59) | 29.13 (1.74) | 29.1 (2.23)
Duration of menses [Mean (Standard Deviation); unit: days] | 5.03 (1.32) | 5.22 (1.28) | 5.11 (1.29)
Type of menstrual pain [Count of Participants; unit: Participants]
  Oppressive-like | 6 | 7 | 13
  Colic-like | 18 | 12 | 30
  Mixed | 5 | 4 | 9
First ever menstrual pain [Count of Participants; unit: Participants]
  1-2 years after menarche | 14 | 7 | 21
  At the time of menarche | 9 | 6 | 15
  1-6 months after menarche | 2 | 8 | 10
  6-12 months after menarche | 3 | 1 | 4
  Other | 1 | 1 | 2
Menstrual pain onset [Count of Participants; unit: Participants]
  Same day | 14 | 6 | 20
  24 hours after | 8 | 5 | 13
  Less than 24 hours before | 3 | 6 | 9
  48-24 hours before | 1 | 6 | 7
  Other | 3 | 0 | 3
Menstrual pain duration [Count of Participants; unit: Participants]
  10-24 hours | 11 | 7 | 18
  24-48 hours | 9 | 6 | 15
  Less than 10 hours | 5 | 7 | 12
  48-72 hours | 3 | 2 | 5
  Other | 1 | 1 | 2
Analgesic used on last menstrual period [Count of Participants; unit: Participants]
  Yes | 12 | 17 | 29
  No | 17 | 6 | 23
Non-pharmacologic treatment used in last menstrual period [Count of Participants; unit: Participants]
  Yes | 10 | 11 | 21
  No | 19 | 12 | 31
Usual menstrual pain - Visual Analogue Scale (VAS1) [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to indicate their usual menstrual pain in a Visual Analogue Scale ranging 0 cm (no pain at al) to 10 cm (worst pain ever)
  units on a scale | 6.34 (1.69) | 6.76 (1.77) | 6.549 (1.71)
Analgesia 1 [Count of Participants; unit: Participants] — Patient were asked if they wanted to use any analgesic prior to the starting the study intervention (no analgesic given)
  Participants
    Yes | 12 | 11 | 23
    No | 17 | 12 | 29
Pain pre-intervention - Visual Analogue Scale (VAS2) [Mean (Standard Deviation); unit: units on a scale] — Patient's were asked to rate their pain immediately prior to starting their allocated intervention using a Visual Analogue Scale ranging 0 cm (no pain at al) to 10 cm (worst pain ever)
  units on a scale | 4.82 (2.04) | 4.97 (1.9) | 4.887 (2.205)
Anxiety (A1) - Abbreviated Zung anxiety scale [Mean (Standard Deviation); unit: units on a scale] — Patients completed the abbreviated Zung anxiety scale in spanish immediately before receiving the allocated intervention. The scale has a total of 10 questions with 4 possible answers "never", "some times", "often", and "always". Each question will have a score of minimum 0 and maximum 3. The final score ranges between 0 and 30.
  units on a scale | 1.8 (0.37) | 1.9 (0.44) | 1.86 (0.38)
Hours with pain [Mean (Standard Deviation); unit: hours] — Patient were asked how many hours they have had their current menstrual pain immediately before receiving the allocated intervention
  hours | 6.27 (5.84) | 6 (5.04) | 6.15 (5.44)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Obtained immediately prior to receiving the allocated intervention Population: Measured pressures in one patient of the silence group was deleted by mistake. Only the measure prior to receiving the intervention were deleted
  mmHg
    number analyzed (Participants) | 29 | 22 | 51
    (all) | 108.97 (11.98) | 105.59 (10.97) | 107.51 (11.56)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Obtained immediately before receiving allocated intervention Population: Measured pressures in one patient of the silence group was deleted by mistake. Only the measure prior to receiving the intervention were deleted
  mmHg
    number analyzed (Participants) | 29 | 22 | 51
    (all) | 71.1 (10.79) | 68.14 (9.88) | 69.82 (10.41)
Mean arterial blood pressure [Mean (Standard Deviation); unit: mmHg] — Obtained immediately prior to receiving the allocated intervention Population: Measured pressures in one patient of the silence group was deleted by mistake. Only the measure prior to receiving the intervention were deleted
  mmHg
    number analyzed (Participants) | 29 | 22 | 51
    (all) | 83.83 (10.32) | 80.62 (9.31) | 82.39 (9.96)
Heart rate [Mean (Standard Deviation); unit: bpm] — Obtained immediately prior to receiving the allocated intervention Population: Measured heart rate in one patient of the silence group was deleted by mistake. Only the measure prior to receiving the intervention was deleted
  bpm
    number analyzed (Participants) | 29 | 22 | 51
    (all) | 75.48 (12.56) | 75.68 (11.87) | 75.62 (12.16)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain From 1-5 Minutes Before (Baseline) to 1- 5 Minutes After the Intervention
Description: Pain scores were measured using a visual analogue scale (VAS) of 10 cm (0 no pain at all, and 10 the worst possible pain) at each time point. Main outcome was calculated from the difference between visual analogue score at 1-5 minutes after (VAS3) minus visual analogue score at 1-5 minutes before the intervention (VAS2).
Time Frame: From 1-5 minutes before the intervention (baseline) to 1-5 minutes after the intervention.
Population: Intention to treat analysis used
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
cm | -1.85 (1.78) | -0.18 (1.8)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Superiority; p = 0.002, t-test, 2 sided

2. Secondary Outcome: Usual Pain Associated to Menses
Description: Mean pain scores measured with a 10 cm visual analogue scale (VAS) where 0 was no pain at all and 10 the worst possible pain. Usual pain was evaluated before the intervention and was known as VAS 1.
Time Frame: 5-10 minutes before the intervention.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
cm | 6.34 (1.69) | 6.76 (1.77)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Equivalence — Equivalence analysis was performed according to pre-defined significant difference of p < 0.01; p = 0.392, t-test, 2 sided

3. Secondary Outcome: Actual Pain 1-5 Minutes Before the Intervention (Baseline).
Description: Mean pain scores measured with a 10 cm visual analogue scale (VAS) where 0 was no pain at all and 10 the worst possible pain. Actual pain was evaluated immediately before the intervention and was known as VAS 2.
Time Frame: 1-5 minutes before the intervention.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
cm | 4.82 (2.04) | 4.97 (2.44)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Equivalence — Equivalence analysis was performed according to pre-defined significant difference of p < 0.01; p = 0.802, t-test, 2 sided

4. Secondary Outcome: Actual Pain 1-5 Minutes After the Intervention.
Description: Mean pain scores measured with a 10 cm visual analogue scale (VAS) where 0 was no pain at all and 10 the worst possible pain. Actual pain was evaluated immediately after the intervention was completed, and was known as VAS 3.
Time Frame: 1-5 minutes after the intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
units on a scale | 2.97 (2.15) | 4.77 (2.68)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Superiority; p = 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Music Group vs Silence Group; Test type: Superiority; p = 0.006, ANCOVA; Fixed factors: group, covariates: pain before (VAS2), age in years, age at menarche, duration of menses, usual pain, anxiety before, hours with pain; Adjusted mean difference = 1.429; Adjusted means: music 3.131 (99% CI 2.62, 3.999) and silence 4.56 (99% CI 3.581, 5.538), F= 8.44, R-square 54.5%

5. Secondary Outcome: Actual Pain 3-6 Hours After the Intervention.
Description: Mean pain scores measured with a 10 cm visual analogue scale (VAS) where 0 was no pain at all and 10 the worst possible pain. Actual pain was evaluated 3-6 hours after the intervention was completed, and was known as VAS 4.
Time Frame: 3-6 hours after the intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 27 | 19
units on a scale | 2.37 (2.31) | 3.63 (2.83)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Superiority; p = 0.11, t-test, 2 sided
Statistical Analysis 2: Comparison: Music Group vs Silence Group; Test type: Superiority; p = 0.370, ANCOVA; Fixed factor: Groups Covariates: Pain before, pain after, age, age menarche, menses duration, usual pain, anxiety before, anxiety after, hours pain; Adjusted mean difference = 0.721 — Adjusted means: music 2.58 (99% CI 1.339, 3.829), and silence 3.305 (1.728, 4.881); F 0.827, R-square 27.2%

6. Secondary Outcome: Anxiety Score Before the Intervention
Description: Using a validated short spanish version of the Zung anxiety scale, anxiety was measured before the intervention. The scale was composed of 10 items. Each item had a 4 Likert point scale (0= never, 1= some times, 2= most of the time, and 3 = always). Final scores ranged from 0, minimum anxiety, and 30 maximum anxiety.
Time Frame: 1-5 minutes before the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
score on a scale | 1.8 (0.37) | 1.9 (0.44)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Equivalence — Equivalence between groups was pre-defined as p > 0.01; p = 0.377, t-test, 2 sided

7. Secondary Outcome: Anxiety Score After the Intervention
Description: Using a validated short spanish version of the Zung anxiety scale, anxiety was measured after the intervention. The scale was composed of 10 items. Each item had a 4 Likert point scale (1= never, 2= some times, 3= most of the time, and 4 = always). Scores ranged from 10, minimum anxiety, and 40 maximum anxiety. For analysis, mean quantitative scores were obtained so 1 was equivalent to minimum anxiety, and 4 to maximum anxiety.
Time Frame: 1-5 minutes after the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
score on a scale | 1.53 (0.33) | 1.73 (0.38)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Superiority; p = 0.049, t-test, 2 sided

8. Secondary Outcome: Anxiety Score 3-6 Hours After the Intervention
Description: Using a validated short spanish version of the Zung anxiety scale, anxiety was measured 3-6 hours after the intervention. The scale was composed of 10 items. Each item had a 4 Likert point scale (0= never, 1= some times, 2= most of the time, and 3= always). Scores ranged from 0, minimum anxiety, and 30 maximum anxiety.
Time Frame: 3-6 hours after fter the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 27 | 19
score on a scale | 1.49 (0.29) | 1.62 (0.36)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Superiority; p = 0.168, t-test, 2 sided

9. Secondary Outcome: Analgesic Requirements Before
Description: Before the intervention patients were asked if they wanted to use any analgesic drug or do any kind of analgesic strategy. Patients simply answered yes or no.
Time Frame: 1-5 minutes before the intervention the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
Participants
  Yes | 12 | 11
  No | 17 | 12
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Equivalence — Equivalence between groups was pre-defined as p > 0.01; p = 0.642, Chi-squared

10. Secondary Outcome: Analgesic Requirements After
Description: After the intervention patients were asked if they wanted to use any analgesic drug or do any kind of analgesic strategy. Patients simply answered yes or no.
Time Frame: 1-5 minutes after the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
Participants
  Yes | 4 | 10
  No | 25 | 13
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Superiority; p = 0.02, Chi-squared

11. Secondary Outcome: Analgesic Use During a Period of 3-6 Hours After the Intervention.
Description: After the intervention, all patients had to register all analgesic drugs (e.g. ibuprofen) or strategy (e.g. local heat) that were used until last pain measurement (VAS 4, 3-6 hours after the intervention).
Time Frame: 3-6 hours after the intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 27 | 19
Participants
  Yes | 6 | 11
  No | 21 | 8
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Superiority; p = 0.025, Chi-squared

12. Secondary Outcome: Systolic Blood Pressure Before the Intervention
Description: Systolic blood pressure in mmHg measured with a calibrated digital sphygmomanometer before the intervention.
Time Frame: 1-5 minutes before the intervention.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
mmHg | 108.97 (11.98) | 105.59 (10.97)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Equivalence — Equivalence between groups determined by pre-deined p > 0.01; p = 0.307, t-test, 2 sided

13. Secondary Outcome: Diastolic Blood Pressure Before the Intervention
Description: Diastolic blood pressure in mmHg measured with a calibrated digital sphygmomanometer before the intervention.
Time Frame: 1-5 minutes before the intervention.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
mmHg | 71.1 (10.79) | 68.14 (9.88)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Equivalence — Equivalence between groups determined by pre-deined p > 0.01; p = 0.318, t-test, 2 sided

14. Secondary Outcome: Heart Rate Before the Intervention
Description: Heart rate measured in beats per minute (bpm) with a calibrated digital sphygmomanometer before the intervention.
Time Frame: 1-5 minutes before the intervention.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
bpm | 75.48 (12.56) | 75.68 (11.87)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Equivalence — Equivalence between groups determined by pre-deined p > 0.01; p = 0.954, t-test, 2 sided

15. Secondary Outcome: Mean Blood Pressure Before the Intervention
Description: Mean blood pressure in mmHg measured with a calibrated digital sphygmomanometer before the intervention.
Time Frame: 1-5 minutes before the intervention.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
mmHg | 83.83 (10.32) | 80.62 (75.68)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Equivalence — Equivalence between groups determined by pre-deined p > 0.01; p = 0.258, t-test, 2 sided

16. Secondary Outcome: Systolic Blood Pressure After the Intervention
Description: Systolic blood pressure in mmHg measured with a calibrated digital sphygmomanometer after the intervention.
Time Frame: 1-5 minutes after the intervention.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
mmHg | 109.66 (14.04) | 103.26 (9.66)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Superiority; p = 0.058, t-test, 2 sided

17. Secondary Outcome: Diastolic Blood Pressure After the Intervention
Description: Diastolic blood pressure in mmHg measured with a calibrated digital sphygmomanometer after the intervention.
Time Frame: 1-5 minutes after the intervention.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
mmHg | 69.9 (9.39) | 65.26 (7.19)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Superiority; p = 0.056, t-test, 2 sided

18. Secondary Outcome: Heart Rate After the Intervention
Description: Heart rate in beats per minute (bpm) measured with a calibrated digital sphygmomanometer after the intervention.
Time Frame: 1-5 minutes after the intervention.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
bpm | 74.48 (11.22) | 74.96 (12.32)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Superiority; p = 0.885, t-test, 2 sided

19. Secondary Outcome: Mean Blood Pressure After the Intervention
Description: Mean blood pressure in mmHg measured with a calibrated digital sphygmomanometer after the intervention.
Time Frame: 1-5 minutes after the intervention.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Music Group | Silence Group
Number analyzed (Participants) | 29 | 23
mmHg | 83.04 (10.22) | 77.92 (6.77)
Statistical Analysis 1: Comparison: Music Group vs Silence Group; Test type: Superiority; p = 0.036, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Description: This is a non-pharmacological intervention, could be classified as behavior, which does not pose any physical, chemical or other type of harm that could be deadly.
Arm/Group | Music Group | Silence Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/23
Other Adverse Events (participants affected / at risk) | 0/29 | 0/23

LIMITATIONS AND CAVEATS:
Patient was not blinded given it is impossible to blind someone from listening to music.

Early termination leading to smaller number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT03593850/Prot_SAP_000.pdf